CLINICAL TRIAL: NCT03186625
Title: Impact of Traditional Chinese Medicine on the Gut Microbiota-dependent Trimethylamine N-oxide in Acute Coronary Syndromes : A Randomized Placebo Controlled Trial
Brief Title: Impact of Traditional Chinese Medicine on the Gut Microbiota-dependent Trimethylamine N-oxide
Acronym: TCM-TMAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: Beijing Genomics Institute (Other)
Responsible Party: Principal Investigator, Lei Wang, Associate Chief Physician, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YN2015MS21
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; gut microbiota; Trimethylamine N-oxide; percutaneous coronary intervention
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compound Panax Notoginseng Granule (Experimental): On the basis of the standard treatment for ACS,eligible participants are randomized to receive Compound Panax Notoginseng Granule when they enroll.
  Interventions: Drug: Compound Panax Notoginseng Granule
- Placebo Granule (Placebo Comparator): On the basis of the standard treatment for ACS,eligible participants are randomized to receive Placebo Granule when they enroll.
  Interventions: Drug: Placebo Granule

INTERVENTIONS:
Drug: Compound Panax Notoginseng Granule — Dosage form:granule. Composition: Panax notoginseng,Codonopsis pilosula,Salvia miltiorrhiza,Pinellia ternata,Medicated Leaven,Coptis chinensis,Citrus reticulata Blanco,etc.
  Frequency:two times a day, one package per time. Duration:three months.
  Arms: Compound Panax Notoginseng Granule
Drug: Placebo Granule — Placebo granule has the same as Compound Panax Notoginseng Granule in the appearance, shape,colour,taste,frequency and duration.
  Arms: Placebo Granule

SUMMARY:
Recent studies highlight the participation of gut microbes in the pathogenesis of both atherosclerotic heart disease and its adverse thrombotic events. Trimethylamine N-oxide (TMAO) is a plasma metabolite shown to be formed through a metaorganismal pathway involving nutrient precursors abundant in a Western diet and the sequential action of gut microbiota. Numerous studies reveal an association between systemic TMAO levels and cardiovascular risks in a variety of stable cohorts. The purpose of this study is to evaluate the efficacy of traditional Chinese Medicine formular (Compound pseudo-ginseng granules ) on the level of TMAO for the patient with acute coronary syndrome(ACS) undergoing percutaneous coronary intervention. 80 patients with ACS would be randomly allocated into interventional group(IG) and control group(CG). The patients in the IG would be administered by oral Compound pseudo-ginseng granules (twice per day ) for 90 days and those in the CG would receive the placebo twice per day during the same period. All of subjects would be administered with standard therapy in accordance with AHA/ACC guideline for ST-elevation myocardial infarction(STEMI) and Non ST-elevation myocardial infarction(NSTEMI).The primary endpoint is the plasma level of TMAO at 90-day follow-up. The second endpoint is the level of lipid, score of The Seattle Angina, fecal DNA extraction and pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

1. acute coronary syndrome (ACS), including ST segment elevate myocardial infarction(STEMI), Non-ST-segment elevation myocardial infarction(NSTEMI) and unstable angina(UA).
2. TCM syndrome: Intermingled Phlegm and Blood Stasis.
3. Aged 18 to 80 years old.
4. sign a consent form.

Exclusion Criteria:

1. Cardiogenic shock.
2. Serious heart failure (NYHA IV or LVEF < 40%).
3. With severe valvular heart disease.
4. Severe hepatic or renal insufficiency, with serum Alanine aminotransferase ( ALT) 3 times higher than normal ceiling or serum creatinine not lower than 265 μmol/L.
5. With acute cerebrovascular disease or severe mental illness.
6. With active bleeding or severe hematopoietic system disease.
7. With malignant tumor or life expectancy in less than three years.
8. Pregnancy or ready to pregnant women, nursing mothers.
9. History of taking antibiotics within the past two months.
10. Participating in other clinical subjects .
11. Failure to sign a consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
the plasma level of TMAO | baseline
  Trimethylamine-N-Oxide(μM) is relative to the prognostic of ACS.
the plasma level of TMAO | 90-days post-procedure
  Trimethylamine-N-Oxide(μM) is relative to the prognostic of ACS.

SECONDARY OUTCOMES:
metagenomic DNA sequencing analysis of faecal microbiome | baseline
  high-throughput sequencing and big data analytics
metagenomic DNA sequencing analysis of faecal microbiome | 90-days post-procedure
  high-throughput sequencing and big data analytics
major adverse cardiac event | 90-days post-procedure
  frequency of the reported cardiovascular events (defined as death, non fatal myocardial infarction,target vessel revascularization and stent thrombosis )
cardiac function | baseline
  left ventricular ejection fraction(LVEF) evaluated by echo
cardiac function | 90-day at follow-up
  left ventricular ejection fraction(LVEF) evaluated by echo
Seattle Angina Questionnaire score | 90-days
  The Seattle Angina Questionnaire is a valid and reliable instrument that measures five clinically important dimensions of health in patients with coronary artery disease (physical limitation, anginal stability, anginal frequency, treatment satisfaction, and disease perception).
The traditional Chinese medicine syndrome scale | change from baseline at 90-days
  The score of phlegm and of blood stasis syndromes is evaluated by Phlegm and blood stasis syndrome questionnaire.
lipid metabolism | change from baseline at 90-days
  low-density lipoprote in cholesterol in mmol/L
lipid metabolism | change from baseline at 90-days
  total cholesterol in cholesterol in mmol/L
inflammatory factors | change from baseline at 90-days
  C-reactive protein in mg/L
platelet function | change from Baseline at 90-days
  maximal aggregation rate of platelet in percent
cardiac biomarkers of necrosis | Change from Baseline at 5 days
  cardiac troponin T (cTnT) in ug/L

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Li, Master, Study Director — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China